CLINICAL TRIAL: NCT01628029
Title: Multimodal Therapy for the Treatment of Sleep Disturbance in Patients With Cancer
Brief Title: Cognitive Behavioral Therapy and Multimodal Therapy in Treating Sleep Disturbance in Patients With Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2012-0120; NCI-2012-01352 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2012-0120 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2012-06-22; First posted 2012-06-26 (Estimated); Results first posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm; Sleep Disorder
MeSH Terms: conditions — Hematologic Neoplasms; Sleep Wake Disorders | interventions — Counseling; Methylphenidate; Phototherapy; Ultraviolet Therapy; Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Arm I (methylphenidate, melatonin, light therapy, CBT) (Experimental): Patients undergo CBT comprising 3 30-minute counseling sessions between baseline and day 14. Patients also receive methylphenidate hydrochloride PO BID and therapeutic melatonin PO QD, and undergo light therapy over 30 minutes for 15 days.
  Interventions: Other: Counseling; Drug: Methylphenidate Hydrochloride; Procedure: Phototherapy; Other: Quality-of-Life Assessment; Drug: Therapeutic Melatonin
- Arm II (placebo, placebo, sham light therapy, CBT) (Experimental): Patients undergo CBT as in Arm I. Patients also receive methylphenidate placebo PO BID and melatonin placebo PO QD, and undergo sham light therapy over 30 minutes for 15 days.
  Interventions: Other: Counseling; Other: Placebo Administration; Other: Quality-of-Life Assessment; Procedure: Sham Intervention
- Arm III (methylphenidate, melatonin, sham light therapy, CBT) (Experimental): Patients undergo CBT as in Arm I. Patients also receive methylphenidate hydrochloride PO BID and therapeutic melatonin PO QD, and undergo sham light therapy over 30 minutes for 15 days.
  Interventions: Other: Counseling; Drug: Methylphenidate Hydrochloride; Other: Quality-of-Life Assessment; Procedure: Sham Intervention; Drug: Therapeutic Melatonin
- Arm IV (methylphenidate, placebo, light therapy, CBT) (Experimental): Patients undergo CBT as in Arm I. Patients also receive methylphenidate hydrochloride PO BID and melatonin placebo PO QD, and undergo light therapy over 30 minutes for 15 days.
  Interventions: Other: Counseling; Drug: Methylphenidate Hydrochloride; Procedure: Phototherapy; Other: Placebo Administration; Other: Quality-of-Life Assessment
- Arm V (placebo, melatonin, light therapy, CBT) (Experimental): Patients undergo CBT as in Arm I. Patients also receive methylphenidate placebo PO BID and therapeutic melatonin PO QD, and undergo light therapy over 30 minutes for 15 days.
  Interventions: Other: Counseling; Procedure: Phototherapy; Other: Placebo Administration; Other: Quality-of-Life Assessment; Drug: Therapeutic Melatonin
- Arm VI (placebo, placebo, light therapy, CBT) (Experimental): Patients undergo CBT as in Arm I. Patients also receive methylphenidate placebo PO BID and melatonin placebo PO QD, and undergo light therapy over 30 minutes for 15 days.
  Interventions: Other: Counseling; Procedure: Phototherapy; Other: Placebo Administration; Other: Quality-of-Life Assessment
- Arm VII (methylphenidate, placebo, sham light therapy, CBT) (Experimental): Patients undergo CBT as in Arm I. Patients also receive methylphenidate hydrochloride PO BID and melatonin placebo PO QD, and undergo sham light therapy over 30 minutes for 15 days.
  Interventions: Other: Counseling; Drug: Methylphenidate Hydrochloride; Other: Placebo Administration; Other: Quality-of-Life Assessment; Procedure: Sham Intervention
- Arm VIII (placebo, melatonin, sham light intervention, CBT) (Experimental): Patients undergo CBT as in Arm I. Patients also receive methylphenidate placebo PO BID and therapeutic melatonin PO QD, and undergo sham light therapy over 30 minutes for 15 days.
  Interventions: Other: Counseling; Other: Placebo Administration; Other: Quality-of-Life Assessment; Procedure: Sham Intervention; Drug: Therapeutic Melatonin

INTERVENTIONS:
Other: Counseling — Undergo CBT
  Other Names: Counseling Intervention
Drug: Methylphenidate Hydrochloride — Given PO
  Other Names: Concerta; Quillivant XR; Ritalin
  Arms: Arm I (methylphenidate, melatonin, light therapy, CBT); Arm III (methylphenidate, melatonin, sham light therapy, CBT); Arm IV (methylphenidate, placebo, light therapy, CBT); Arm VII (methylphenidate, placebo, sham light therapy, CBT)
Procedure: Phototherapy — Undergo light therapy
  Other Names: Actinotherapy; Bright Light Therapy; light therapy
  Arms: Arm I (methylphenidate, melatonin, light therapy, CBT); Arm IV (methylphenidate, placebo, light therapy, CBT); Arm V (placebo, melatonin, light therapy, CBT); Arm VI (placebo, placebo, light therapy, CBT)
Other: Placebo Administration — Given PO
  Arms: Arm II (placebo, placebo, sham light therapy, CBT); Arm IV (methylphenidate, placebo, light therapy, CBT); Arm V (placebo, melatonin, light therapy, CBT); Arm VI (placebo, placebo, light therapy, CBT); Arm VII (methylphenidate, placebo, sham light therapy, CBT); Arm VIII (placebo, melatonin, sham light intervention, CBT)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Procedure: Sham Intervention — Undergo sham light therapy
  Other Names: Sham Comparator
  Arms: Arm II (placebo, placebo, sham light therapy, CBT); Arm III (methylphenidate, melatonin, sham light therapy, CBT); Arm VII (methylphenidate, placebo, sham light therapy, CBT); Arm VIII (placebo, melatonin, sham light intervention, CBT)
Drug: Therapeutic Melatonin — Given PO
  Other Names: Circadin; Melatonin; Melaxen
  Arms: Arm I (methylphenidate, melatonin, light therapy, CBT); Arm III (methylphenidate, melatonin, sham light therapy, CBT); Arm V (placebo, melatonin, light therapy, CBT); Arm VIII (placebo, melatonin, sham light intervention, CBT)

SUMMARY:
This randomized phase II trial studies how well cognitive behavioral therapy and multimodal therapy works in treating sleep disturbance in patients with cancer. Cognitive behavioral therapy may help reduce sleep disturbances, fatigue, and insomnia as well as improve the well-being and quality of life of patients with cancer when given together with methylphenidate hydrochloride, therapeutic melatonin, and light therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To obtain preliminary estimates of the effects of cognitive behavioral therapy (CBT) and various treatments (light therapy, melatonin, methylphenidate [methylphenidate hydrochloride]) and combinations of treatments in multimodal therapy (MMT) in reducing sleep disturbance in patients with cancer, as measured by change in Pittsburgh Sleep Quality Index (PSQI) scores taken at baseline and on day 15.

SECONDARY OBJECTIVES:

I. To explore the effect of MMT on Insomnia Severity Index, cancer related symptoms (fatigue [Functional Assessment of Chronic Illness Therapy (FACIT-F) subscale, Edmonton Symptom Assessment System (ESAS)], anxiety, depression anxiety [Hospital Anxiety Depression Scale (HADS), ESAS]), quality of life (Functional Assessment of Cancer Therapy-General [FACT-G], ESAS), and physical activity/sleep efficacy (actigraphy), before and after treatment with various sleep disturbance (SD) treatment combinations of MMT.

II. To determine the safety of MMT (type, frequency, and severity of the adverse events).

OUTLINE: Patients are randomized to 1 of 8 treatment arms.

ARM I: Patients undergo CBT comprising 3 30-minute counseling sessions between baseline and day 14. Patients also receive methylphenidate hydrochloride orally (PO) twice daily (BID) and therapeutic melatonin PO once daily (QD), and undergo light therapy over 30 minutes for 15 days.

ARM II: Patients undergo CBT as in Arm I. Patients also receive methylphenidate placebo PO BID and melatonin placebo PO QD, and undergo sham light therapy over 30 minutes for 15 days.

ARM III: Patients undergo CBT as in Arm I. Patients also receive methylphenidate hydrochloride PO BID and therapeutic melatonin PO QD, and undergo sham light therapy over 30 minutes for 15 days.

ARM IV: Patients undergo CBT as in Arm I. Patients also receive methylphenidate hydrochloride PO BID and melatonin placebo PO QD, and undergo light therapy over 30 minutes for 15 days.

ARM V: Patients undergo CBT as in Arm I. Patients also receive methylphenidate placebo PO BID and therapeutic melatonin PO QD, and undergo light therapy over 30 minutes for 15 days.

ARM VI: Patients undergo CBT as in Arm I. Patients also receive methylphenidate placebo PO BID and melatonin placebo PO QD, and undergo light therapy over 30 minutes for 15 days.

ARM VII: Patients undergo CBT as in Arm I. Patients also receive methylphenidate hydrochloride PO BID and melatonin placebo PO QD, and undergo sham light therapy over 30 minutes for 15 days.

ARM VIII: Patients undergo CBT as in Arm I. Patients also receive methylphenidate placebo PO BID and therapeutic melatonin PO QD, and undergo sham light therapy over 30 minutes for 15 days.

Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up on days 29 and 45.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients currently on cancer therapy with a positive screening for SD (screening PSQI score >= 5)
* Patients should have a Zubrod =< 2
* Patients with no pain and with stable pain (defined as pain under control and on stable doses of opioids for 1 week) are eligible
* Memorial delirium assessment scale =< 13
* Controlled pain and depression symptoms, if present (defined as no change in the morphine equivalent dose of 30% or change in the dose of antidepressant medication in the past 2 weeks)
* All patients who are receiving chemotherapy and/or radiation therapy are eligible for study if they have completed > 1 week of radiation therapy, and if they have been approved to go on study by their primary oncologist; the principal investigator (PI)/designated research staff of this study will obtain and document approval from the primary oncologist and principal investigator of the clinical trial in case the patient is on another clinical trial as referenced in the patient's study documents
* Serum creatinine =< 2.0 mg/dL
* Total bilirubin =< 1.5 mg/dL
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2 x upper limit of normal (ULN) or =< 5 x ULN if hepatic metastases are present
* Patients on stable doses (defined as same dose for 2 weeks) of dexamethasone, mirtazapine, zolpidem, benzodiazepines, phenothiazines are allowed to participate in the study

Exclusion Criteria:

* Have a major contraindication to methylphenidate (MP) (e.g., allergy/hypersensitivity to study medications or their constituents), light therapy (e.g., currently receiving ultraviolet A [UVA]/ultraviolet B [UVB] therapy), cognitive behavioral therapy (e.g., schizophrenia), or conditions making adherence difficult as determined by the attending physician
* Currently taking MP or have taken it within the previous 10 days
* Patients with a diagnosis of polysomnographically confirmed obstructive sleep apnea or narcolepsy
* Regularly used cognitive behavioral therapy in the last 6 weeks for sleep disturbance
* Unable to complete the baseline assessment forms or to understand the recommendations for participation in the study
* Currently with a diagnosis of major depression, manic depressive disorder, obsessive-compulsive disorder, or schizophrenia)
* Need monoamine oxidase inhibitors, tricyclic antidepressants, or clonidine
* Have glaucoma
* Symptomatic tachycardia and uncontrolled hypertension (determined to be clinically significant by the PI)
* Currently receiving anticonvulsants (phenobarbital, diphenylhydantoin, primidone), phenylbutazone, clonidine, and/or tricyclic drugs (imipramine, clomipramine, or desipramine)
* Unable to speak and understand English
* Persons with congenital blindness and self-reported acquired blindness (independent of the cause) with no light perception
* Patients with a history of retinal disease
* Patients with > 2 hours of direct exposure to outdoor natural light per day by interview with the Study Coordinator
* Patients with a diagnosis of obesity hypoventilation syndrome
* Positive pregnancy test for women of childbearing potential, as defined by intact uterus and ovaries, and a history of menses within the last 12 months; pregnancy test to be performed no greater than 14 days prior to consent in study; in cases of women with elevated beta (b)-human chorionic gonadotropin (HCG), these candidates will be eligible to participate so long as the level of b-HCG is not consistent with pregnancy; women of childbearing potential need to be on or use contraception, or be abstinent during the study period; their male partners must also use contraception (condom) or maintain abstinence; birth control specifications: women who are able to become pregnant must use birth control during the study and for 30 days after
* Women who are nursing
* Patients who have taken melatonin within the past two weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2014-01-15 (Actual); Primary Completion 2025-12-22 (Actual); Study Completion 2028-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sriram Yennu, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Yennurajalingam S, Carmack C, Balachandran D, Eng C, Lim B, Delgado M, Guzman Gutierrez D, Raznahan M, Park M, Hess KR, Williams JL, Lu Z, Ochoa J, Bruera E. Sleep disturbance in patients with cancer: a feasibility study of multimodal therapy. BMJ Support Palliat Care. 2021 Jun;11(2):170-179. doi: 10.1136/bmjspcare-2019-001877. Epub 2020 Jan 10. PMID 31924662
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Dim Red Light + Placebo + Placebo: 50 lux once a day (30 minutes) for 14 days + Melatonin Placebo + Methylphenidate Placebo
- Bright White Light Therpay + Melatonin + Placebo: 1350 lux once a day (30 minutes) for 14 days + Melatonin 20mg tablet orally at bedtime for 14 days + Methylphenidate Placebo
- Dim Red Light + Melatonin + Methylphenidate: 50 lux once a day (30 minutes) for 14 days + Melatonin 20mg tablet orally at bedtime for 14 days + Methylphenidate 5mg tablet orally twice daily for 14 days
- Bright White Light Therapy + Placebo + Methylphenidate: 1350 lux once a day (30 minutes) for 14 days + Melatonin Placebo + Methylphenidate 5mg tablet orally twice daily for 14 days
- Bright White Light Therapy + Placebo + Placebo: 1350 lux once a day (30 minutes) for 14 days + Melatonin Placebo + Methylphenidate Placebo
- Dim Red Light + Melatonin + Placebo: 50 lux once a day (30 minutes) for 14 days + Melatonin 20mg tablet orally at bedtime for 14 days + Methylphenidate Placebo
- Dim Red Light + Placebo + Methylphenidate: 50 lux once a day (30 minutes) for 14 days + Melatonin Placebo + Methylphenidate 5mg tablet orally twice daily for 14 days
- Bright White Light Therapy + Melatonin + Methylphenidate: 1350 lux once a day (30 minutes) for 14 days + Melatonin 20mg tablet orally at bedtime for 14 days + Methylphenidate 5mg tablet orally twice daily for 14 days
Period: Overall Study
Arm/Group | Dim Red Light + Placebo + Placebo | Bright White Light Therpay + Melatonin + Placebo | Dim Red Light + Melatonin + Methylphenidate | Bright White Light Therapy + Placebo + Methylphenidate | Bright White Light Therapy + Placebo + Placebo | Dim Red Light + Melatonin + Placebo | Dim Red Light + Placebo + Methylphenidate | Bright White Light Therapy + Melatonin + Methylphenidate
Started | 9 | 8 | 8 | 9 | 9 | 8 | 7 | 9
Completed | 8 | 6 | 5 | 8 | 8 | 7 | 5 | 7
Not Completed | 1 | 2 | 3 | 1 | 1 | 1 | 2 | 2
Not completed — Symptom burden | 1 | 0 | 1 | 0 | 1 | 1 | 2 | 2
Not completed — Withdrew due to lack of benefit | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Non compliant | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — started different cancer treatment clinical trial | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Incomplete primary outcome assessment | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dim Red Light + Placebo + Placebo | Bright White Light Therpay + Melatonin + Placebo | Dim Red Light + Melatonin + Methylphenidate | Bright White Light Therapy + Placebo + Methylphenidate | Bright White Light Therapy + Placebo + Placebo | Dim Red Light + Melatonin + Placebo | Dim Red Light + Placebo + Methylphenidate | Bright White Light Therapy + Melatonin + Methylphenidate | Total
Number analyzed (Participants) | 9 | 6 | 7 | 9 | 9 | 8 | 7 | 9 | 64
Age, Continuous [Median (Full Range); unit: years] | 54 [38 to 63] | 54 [34 to 74] | 50 [41 to 65] | 54 [34 to 73] | 57 [40 to 66] | 55 [27 to 71] | 43 [24 to 57] | 55 [31 to 68] | 52.5 [24 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 3 | 6 | 7 | 4 | 4 | 4 | 42
  Male | 1 | 0 | 4 | 3 | 2 | 4 | 3 | 5 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 1 | 1 | 1 | 3 | 0 | 1 | 10
  Not Hispanic or Latino | 8 | 4 | 6 | 8 | 8 | 5 | 7 | 8 | 54
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 1 | 1 | 2 | 2 | 2 | 10
  White | 7 | 6 | 5 | 7 | 7 | 6 | 5 | 7 | 50
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 6 | 7 | 9 | 9 | 8 | 7 | 9 | 64
Cancer Distribution of the participants [Count of Participants; unit: Participants]
  GI | 2 | 0 | 2 | 2 | 3 | 2 | 4 | 1 | 16
  GU | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 6
  Breast | 4 | 3 | 2 | 5 | 1 | 1 | 1 | 2 | 19
  GYN | 2 | 0 | 0 | 0 | 4 | 1 | 0 | 1 | 8
  Lung | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 6
  Sarcoma | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 5
  Other | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Pittsburgh Sleep Quality Index (PSQI) Score Change
Description: PSQI consists of 19 items, and it measures several different aspects of sleep, offering seven component scores and one composite score. The component scores consist of subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Each component score ranges from 0 (no difficulty/good) to 3 (severe difficulty/poor). The global PSQI score is then calculated by totaling (summed) seven component scores, providing an overall score ranging from 0 to 21, where 0 indicates very good sleep quality and 21 signifies very poor sleep quality. A global score of greater than 5 often suggests significant sleep problems. In this study, Wilcoxon signed-rank test was used to determine the p value.
Time Frame: Baseline and Day 15
Population: Those who completed the study assessment and treatment
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Dim Red Light + Placebo + Placebo | Bright White Light Therpay + Melatonin + Placebo | Dim Red Light + Melatonin + Methylphenidate | Bright White Light Therapy + Placebo + Methylphenidate | Bright White Light Therapy + Placebo + Placebo | Dim Red Light + Melatonin + Placebo | Dim Red Light + Placebo + Methylphenidate | Bright White Light Therapy + Melatonin + Methylphenidate
Number analyzed (Participants) | 8 | 6 | 5 | 8 | 8 | 7 | 5 | 7
score on a scale | -1.5 [-5.0 to 0.0] | -6.5 [-8.0 to -4.0] | -1.0 [-5.0 to 0.0] | -3.0 [-6.0 to 1.5] | -3.0 [-8.0 to -1.0] | -2.0 [-5.0 to 2.0] | -3.0 [-3.0 to -2.0] | -5.0 [-7.0 to -2.0]

2. Secondary Outcome: Functional Assessment of Chronic Illness Therapy- Fatigue (FACIT-F) Subscale Score Change
Description: There are 13 items in this FACIT-F subscale. In this subscale, the patient rates the intensity of fatigue and its related symptoms on a scale from 0 to 4 in the past week. The total score can range between 0 and 52, with higher scores denoting less fatigue. Wilcoxon signed-rank test was used to determine the p-value.
Time Frame: Baseline and Day 15
Population: Those who completed the study assessment and treatment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Dim Red Light + Placebo + Placebo | Bright White Light Therpay + Melatonin + Placebo | Dim Red Light + Melatonin + Methylphenidate | Bright White Light Therapy + Placebo + Methylphenidate | Bright White Light Therapy + Placebo + Placebo | Dim Red Light + Melatonin + Placebo | Dim Red Light + Placebo + Methylphenidate | Bright White Light Therapy + Melatonin + Methylphenidate
Number analyzed (Participants) | 8 | 6 | 5 | 8 | 8 | 7 | 5 | 7
score on a scale | 7.0 [1.5 to 15.0] | 2.5 [-5.0 to 16.0] | 5.0 [-2.0 to 17.0] | 7.0 [5.0 to 10.5] | 1.0 [-8.5 to 13.0] | 13.0 [-4.0 to 14.0] | 11.0 [11.0 to 13.0] | 8.0 [5.0 to 22.0]

3. Secondary Outcome: Insomnia Severity Index (ISI)) Score Change
Description: The ISI is a 7-item questionnaire designed to evaluate insomnia severity. Each item is rated using a 5-point Likert scale ranging from 0 (not at all) to 4 (very much), for a total score ranging from 0 to 28 with a cut-off score of 10 or greater indicating significant insomnia. Wilcoxon signed-rank test was used to determine the p-value.
Time Frame: Baseline and Day 15
Population: Those who completed the study assessment and treatment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Dim Red Light + Placebo + Placebo | Bright White Light Therpay + Melatonin + Placebo | Dim Red Light + Melatonin + Methylphenidate | Bright White Light Therapy + Placebo + Methylphenidate | Bright White Light Therapy + Placebo + Placebo | Dim Red Light + Melatonin + Placebo | Dim Red Light + Placebo + Methylphenidate | Bright White Light Therapy + Melatonin + Methylphenidate
Number analyzed (Participants) | 8 | 6 | 5 | 8 | 8 | 7 | 5 | 7
score on a scale | -6.5 [-9.5 to -2.5] | -11.0 [-13.0 to -3.0] | -10.0 [-12.0 to -7.0] | -4.0 [-9.0 to -2.5] | -9.0 [-13.0 to -6.0] | -4.0 [-6.0 to 1.0] | -13.0 [-14.0 to -1.0] | -7.5 [-13.0 to -4.0]

4. Secondary Outcome: Functional Assessment of Cancer Therapy - General (FACT-G) Score Change
Description: The FACT-G is a quality-of-life instrument that is commonly used in cancer clinical trials. FACT-G consists of 27 general quality-of-life questions divided into 4 domains (physical, social, emotional and functional). The patient rates the intensity of symptoms on a Likert scale from 0 (not at all) to 4 (very much). Total score ranges from 0-108 with higher score indicates better Quality of Life. Wilcoxon signed-rank test was used to determine the p-value.
Time Frame: Baseline and Day 15
Population: Those who completed the study assessment and treatment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Dim Red Light + Placebo + Placebo | Bright White Light Therpay + Melatonin + Placebo | Dim Red Light + Melatonin + Methylphenidate | Bright White Light Therapy + Placebo + Methylphenidate | Bright White Light Therapy + Placebo + Placebo | Dim Red Light + Melatonin + Placebo | Dim Red Light + Placebo + Methylphenidate | Bright White Light Therapy + Melatonin + Methylphenidate
Number analyzed (Participants) | 8 | 6 | 5 | 8 | 8 | 7 | 5 | 7
score on a scale | 4.5 [0.0 to 10.0] | 10.5 [5.0 to 13.0] | 7.0 [6.0 to 19.0] | 11.0 [-5.0 to 11.0] | 12.0 [1.0 to 19.0] | 5.0 [1.0 to 17.0] | 10.0 [7.0 to 25.0] | 3.0 [-1.0 to 11.0]

ADVERSE EVENTS:
Time Frame: Baseline to Day 15
Arm/Group | Dim Red Light + Placebo + Placebo | Bright White Light Therpay + Melatonin + Placebo | Dim Red Light + Melatonin + Methylphenidate | Bright White Light Therapy + Placebo + Methylphenidate | Bright White Light Therapy + Placebo + Placebo | Dim Red Light + Melatonin + Placebo | Dim Red Light + Placebo + Methylphenidate | Bright White Light Therapy + Melatonin + Methylphenidate
All-Cause Mortality (participants affected / at risk) | 1/9 | 0/6 | 0/7 | 0/9 | 0/9 | 0/8 | 0/7 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/6 | 0/7 | 0/9 | 0/9 | 0/8 | 0/7 | 0/9
Other Adverse Events (participants affected / at risk) | 4/9 | 0/6 | 1/7 | 2/9 | 1/9 | 2/8 | 3/7 | 0/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dim Red Light + Placebo + Placebo (N=9) | Bright White Light Therpay + Melatonin + Placebo (N=6) | Dim Red Light + Melatonin + Methylphenidate (N=7) | Bright White Light Therapy + Placebo + Methylphenidate (N=9) | Bright White Light Therapy + Placebo + Placebo (N=9) | Dim Red Light + Melatonin + Placebo (N=8) | Dim Red Light + Placebo + Methylphenidate (N=7) | Bright White Light Therapy + Melatonin + Methylphenidate (N=9)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Death (NOS) (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oedema limbs (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic Infection (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-07): https://cdn.clinicaltrials.gov/large-docs/29/NCT01628029/Prot_SAP_000.pdf